CLINICAL TRIAL: NCT07019181
Title: Tislelizumab Combined With Chemotherapy for the Perioperative Treatment of Esophageal Squamous Carcinoma： Single-arm Clinical Phase II Study
Brief Title: Tislelizumab Combined With Chemotherapy for the Perioperative Treatment of Esophageal Squamous Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-2024KY088-01
Record Dates: First submitted 2025-05-21; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — tislelizumab; Albumin-Bound Paclitaxel; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tislelizumab combined with chemotherapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: albumin-bound paclitaxel; Drug: Nedaplatin

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab, 200mg, intravenously over 30 - 60 minutes, day 1 of every 3 weeks
Drug: albumin-bound paclitaxel — albumin-bound paclitaxel 260mg/m2，day 1 of every 3 weeks
Drug: Nedaplatin — Nedaplatin 80mg/m2，day 1 of every 3 weeks

SUMMARY:
Evaluating the rate of pathologic complete remission in patients with squamous esophageal cancer treated perioperatively with tislelizumab in combination with chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Subjects were enrolled in the study and signed an informed consent form.
* Male or female patients between the ages of 18 and 75.
* Patients with esophageal squamous carcinoma diagnosed by histopathology.
* According to the TNM staging system of esophageal cancer in the 8th edition of the AJCC,the disease is in the stage of cT3-4aN0M0 or cT1b-4aN+M0 (confirmed by thoracic and abdominal enhancement CT/MRI), and the lesion is located in the thoracic segment.
* ECOG score: 0-1.
* Normal functioning of major organs, i.e. meeting the following criteria.

  1. Blood count (no blood transfusions, granulocyte colony-stimulating factor [G-CSF], or other medications corrected within 14 days prior to treatment); and Absolute neutrophil count (ANC) ≥1.5×109/L; hemoglobin (HB) ≥9.0 g/dL; and Platelet count (PLT) ≥ 100 x 109/L;
  2. blood biochemistry Creatinine clearance ≥60 mL/min. Total bilirubin (TBIL) ≤ 1.5 x ULN. Albuminous aminotransferase (AST) or albuminous aminotransferase (ALT) levels ≤ 2.5 x ULN;
* Expected survival > 6 months.
* Female subjects of childbearing potential and male subjects with partners of childbearing potential are required to use a medically approved contraceptive method during study treatment and for at least 6 months after the last treatment.

Exclusion Criteria:

* The presence of clinically uncontrolled chest that required repeated drainage or medical intervention (within 2 weeks prior to randomization) Hydrocele, pericardial hydrocele or ascites;
* Known intolerance or resistance to chemotherapy specified in the trial protocol;
* Have received any other ESCC anti-tumor therapy (e.g., targeting PD-1, PD-L1, PD-L2) Or other tumor immunotherapy, radiotherapy, targeted therapy, ablation, or other systemic or local anti-tumor therapy);
* Patients who have an active autoimmune disease or have a history of an autoimmune disease but may relapse may have a known abnormality History of body organ transplantation or allogeneic hematopoietic stem cell transplantation;
* A history of interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic disease, including pulmonary fibrosis, Acute lung disease;
* There were severe chronic or active patients requiring systemic antimicrobial therapy, antifungal therapy or antiviral therapy before enrollment Infection (including tuberculosis infection, etc.);
* Have a known history of HIV infection;
* The presence of any serious or uncontrolled systemic disease, including but not limited to:

Unstable angina pectoris, congestive heart failure, New York Heart Association (NYHA) grade ≥ 2 chronic heart failure; Any arterial thrombosis, embolism, or ischemia, such as myocardial infarction, cerebrovascular accident, or transient ischemic attack, during the 6 months prior to the first dose of the study; Uncontrolled hypertension (i.e., ≥ CTC-AE level 2 hypertension after medication); active pulmonary tuberculosis; those who have a history of psychotropic substance abuse and cannot abstain or have mental disorders;

* Had other malignancies in the past 5 years (cured skin basal cell carcinoma, breast carcinoma in situ and Except primary cervical cancer);
* Had received live vaccine within 28 days prior to enrollment;
* Have participated in other therapeutic clinical trials within 4 weeks;
* And those deemed unsuitable for inclusion by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | 4 weeks after surgery
  Pathological complete responseTotal tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell

SECONDARY OUTCOMES:
Major pathological response rate | 4 weeks after surgery
  Total/moderate tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell
Objective Response Rate | At the end of Cycle 2(each cycle is 28 days)
  Objective Response Rate Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor